CLINICAL TRIAL: NCT01949051
Title: A Randomized, Double-blind, Placebo Controlled, 3 Way Cross Over Study in Subjects With Allergic Rhinitis to Assess the Effect of Intranasal Repeat Doses of Levocabastine When Administered Once Daily or Twice Daily on the Symptoms of Rhinitis in an Allergen Challenge Chamber
Brief Title: A Study to Assess Intranasal Repeat Dose Effect of Levocabastine in the Subjects With Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200285
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Rhinitis, Allergic, Perennial and Seasonal
Keywords: Allergic rhinitis; levocabastine; allergen challenge
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic | interventions — levocabastine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Levocabastine Arm (Experimental): Subjects will be assigned to one of six treatment sequences (ABC, BCA, CAB, ACB, BAC, CBA) in accordance with the randomisation schedule. A = Two, 50 microgram (mcg) sprays per nostril of levocabastine QD in the morning. Total dose of 200 mcg. Two, 0 mcg sprays from placebo to match vehicle in the evening; B = Two, 50 mcg sprays per nostril of levocabastine BID in the morning and evening. Total dose of 400 mcg; C = Two, 0 mcg sprays per nostril from placebo vehicle in morning and evenings.
  Interventions: Drug: Levocabastine; Drug: Placebo

INTERVENTIONS:
Drug: Levocabastine — Intranasal aqueous 50 mcg microsuspension of levocabastine supplied in an amber glass bottle fitted with a white top actuated plastic metering atomising spray pump filled with a uniform white suspension
Drug: Placebo — Intranasal aqueous 0 mcg microsuspension supplied in an amber glass bottle fitted with a white top actuated plastic metering atomising spray pump filled with a uniform white suspension

SUMMARY:
This study will be a randomized, double blind, placebo controlled, 3-way cross over design in allergic rhinitis subjects. Subjects will receive repeat doses of intra-nasal levocabastine for 7 days in each period and the duration of the study will be about 13 weeks. An Environmental Exposure Chamber (EEC) will be used in this study. The primary objective of the study is to investigate the non-inferiority effect of 7 days treatment with levocabastine on nasal symptoms elicited by an EEC when administered once daily (QD) compared with twice daily (BID). Also study will be conducted to investigate the superiority of effect of 7 days treatment with levocabastine (QD and BID) on nasal symptoms elicited by an EEC in subjects compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Allergic Rhinitis (AR), as determined by the presence of seasonal or perennial rhinitis symptoms for several months per year, for more than 1 year and are not attributed to infections or nasal abnormalities.
* Subjects have a TNSS score of >=6 at the baseline screening allergen challenge. Total nasal symptom score is the sum of nasal congestion, rhinorrhoea, nasal itch and sneeze, each of which are scored on a scale from 0 to 3.
* Subjects have a positive skin prick test (wheal >=4 millimeter [mm]) for seasonal pollen at or within the 12 months preceding the screening visit.
* Subjects have a positive radioallergosorbent test (RAST) (>=class 2) for seasonal pollen at or within the 12 months preceding the screening visit.
* There are no conditions or factors that would make the subject unlikely to be able to stay in the chamber for 4 hours.
* Male/females between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 19 - 30 kg per meter square (m^2) (inclusive).
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy (for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records); or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli international unit per milliliter (MlU/mL) and estradiol <40 picogram (pg)/mL (<147 picomol per liter [pmol/L]) is confirmatory); child-bearing potential with negative pregnancy test as determined by urine human chorionic gonadotropin (hCG) test at screening or prior to dosing and agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 1 week post-last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subjects should be non-smokers, which for this study is defined as having smoked <10 packs per year in their lifetime, and have not smoked in the 6 months prior to the screening visit.
* Alanine aminotransferase (ALT), alkaline phosphatase (ALP) and bilirubin <=1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged corrected QT interval (QTc) values of triplicate electrocardiogram (ECGs) obtained over a brief recording period: Fridericia QTc (QTcF) <450 milliseconds (msec).

Exclusion Criteria:

* Nasal abnormalities likely to affect the outcome of the study, i.e. nasal septal perforation, nasal polyps, sinusitis and other nasal malformations.
* History of frequent nosebleeds.
* Subjects with rhinitis medicamentosa.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Significant renal impairment, which based on the opinion of the investigator, would preclude the subject's participation in the study.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360mL) of beer, 5 ounces (150mL) of wine or 1.5 ounces (45ml) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Chronic oral steroids discontinued less than 6 months prior to screening.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

Subjects who are using some of the medications below on an as needed basis, may participate in the study if they remain free of medication for the following periods of time prior to screening and prior to dosing (study drugs): Nasal antihistamines: 72 hours, Oral antihistamines A (cetirizine, fexofenadine, loratadine, desloratadine): 72 hours, Oral antihistamines B (all others): 72hours, Eye and Nasal Levocasbastine: 7 days, Nasal decongestants: 24 hours, Oral decongestants: 24 hours, Nasal glucocorticosteroids: 7 days, Inhaled glucocorticoids: 1 week, Oral glucocorticosteroids: 12 weeks, Oral leukotriene receptor antagonists: 7 days, Oral 5-lipoxygenase inhibitors: 7 days, Oral methylxanthines: 7 days

* Subjects with recent upper respiratory tract infections (URTIs) will be allowed in the study only if their nasal symptoms associated with the URTI have been completely resolved for more than 3 weeks prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-02-04 (Actual); Study Completion 2014-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Murdoch RD, Bareille P, Ignar D, Mark S, Miller SR, Gupta A, Salapatek AM, Patel P. Once-daily dosing of levocabastine has comparable efficacy to twice-daily dosing in the treatment of allergic rhinitis assessed in an allergen challenge chamber. Int J Clin Pharmacol Ther. 2015 Oct;53(10):811-8. doi: 10.5414/CP202389. PMID 26249767
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 200285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who met the eligibility criteria at Screening were randomized to 1 of 6 treatment sequences. The treatment phase was comprised of three 7-day treatment periods, each separated by a 14- to 20-day washout period.
Groups:
- Sequence 1: Levo 200 µg, Levo 400µg, Placebo: Participants received levocabastine (Levo) 200 micrograms (µg), Levo 400µg and placebo in Treatment Periods 1, 2, and 3, respectively. Participants received the Levo 200 µg once daily (OD) in the morning as 2 nasal sprays (50 µg per spray) and placebo in the evening into each nostril or placebo/ Levo 400 µg twice daily (BID) in the morning and evening as 2 nasal sprays (50 µg per spray) into each nostril for 7 days. The three treatment periods were separated by a washout period of 14 to 20 days.
- Sequence 2: Levo 400µg, Placebo and Levo 200µg: Participants received Levo 400µg, placebo and Levo 200µg in Treatment Periods 1, 2, and 3, respectively. Participants received the Levo 200 µg OD in the morning as 2 nasal sprays (50 µg per spray) and placebo in the evening into each nostril or placebo/ Levo 400 µg BID in the morning and evening as 2 nasal sprays (50 µg per spray) into each nostril for 7 days. The three treatment periods were separated by a washout period of 14 to 20 days.
- Sequence 3: Placebo, Levo 200µg and Levo 400µg: Participants received placebo, Levo 200µg and Levo 400µg in Treatment Periods 1, 2, and 3, respectively. Participants received the Levo 200 µg OD in the morning as 2 nasal sprays (50 µg per spray) and placebo in the evening into each nostril or placebo/ Levo 400 µg BID in the morning and evening as 2 nasal sprays (50 µg per spray) into each nostril for 7 days. The three treatment periods were separated by a washout period of 14 to 20 days.
- Sequence 4: Levo 200µg, Placebo, and Levo 400µg: Participants received Levo 200µg, placebo, and Levo 400µg in Treatment Periods 1, 2, and 3, respectively. Participants received the Levo 200 µg OD in the morning as 2 nasal sprays (50 µg per spray) and placebo in the evening into each nostril or placebo/ Levo 400 µg BID in the morning and evening as 2 nasal sprays (50 µg per spray) into each nostril for 7 days. The three treatment periods were separated by a washout period of 14 to 20 days.
- Sequence 5: Levo 400µg, Levo 200µg and Placebo: Participants received Levo 400µg, Levo 200µg and placebo in Treatment Periods 1, 2, and 3, respectively. Participants received the Levo 200 µg OD in the morning as 2 nasal sprays (50 µg per spray) and placebo in the evening into each nostril or placebo/ Levo 400 µg BID in the morning and evening as 2 nasal sprays (50 µg per spray) into each nostril for 7 days. The three treatment periods were separated by a washout period of 14 to 20 days.
- Sequence 6: Placebo, Levo 400µg and Levo 200µg: Participants received placebo, Levo 400µg and Levo 200µg in Treatment Periods 1, 2, and 3, respectively. Participants received the Levo 200 µg OD in the morning as 2 nasal sprays (50 µg per spray) and placebo in the evening into each nostril or placebo/ Levo 400 µg BID in the morning and evening as 2 nasal sprays (50 µg per spray) into each nostril for 7 days. The three treatment periods were separated by a washout period of 14 to 20 days.
Period: Treatment Period 1 (7 Days)
Arm/Group | Sequence 1: Levo 200 µg, Levo 400µg, Placebo | Sequence 2: Levo 400µg, Placebo and Levo 200µg | Sequence 3: Placebo, Levo 200µg and Levo 400µg | Sequence 4: Levo 200µg, Placebo, and Levo 400µg | Sequence 5: Levo 400µg, Levo 200µg and Placebo | Sequence 6: Placebo, Levo 400µg and Levo 200µg
Started | 13 | 13 | 13 | 13 | 13 | 13
Completed | 11 | 13 | 13 | 12 | 13 | 13
Not Completed | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (14 to 20 Days)
Arm/Group | Sequence 1: Levo 200 µg, Levo 400µg, Placebo | Sequence 2: Levo 400µg, Placebo and Levo 200µg | Sequence 3: Placebo, Levo 200µg and Levo 400µg | Sequence 4: Levo 200µg, Placebo, and Levo 400µg | Sequence 5: Levo 400µg, Levo 200µg and Placebo | Sequence 6: Placebo, Levo 400µg and Levo 200µg
Started | 11 | 13 | 13 | 12 | 13 | 13
Completed | 11 | 13 | 13 | 12 | 13 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (7 Days)
Arm/Group | Sequence 1: Levo 200 µg, Levo 400µg, Placebo | Sequence 2: Levo 400µg, Placebo and Levo 200µg | Sequence 3: Placebo, Levo 200µg and Levo 400µg | Sequence 4: Levo 200µg, Placebo, and Levo 400µg | Sequence 5: Levo 400µg, Levo 200µg and Placebo | Sequence 6: Placebo, Levo 400µg and Levo 200µg
Started | 11 | 13 | 13 | 12 | 13 | 13
Completed | 11 | 12 | 12 | 12 | 13 | 12
Not Completed | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout Period 2 (14 to 20 Days)
Arm/Group | Sequence 1: Levo 200 µg, Levo 400µg, Placebo | Sequence 2: Levo 400µg, Placebo and Levo 200µg | Sequence 3: Placebo, Levo 200µg and Levo 400µg | Sequence 4: Levo 200µg, Placebo, and Levo 400µg | Sequence 5: Levo 400µg, Levo 200µg and Placebo | Sequence 6: Placebo, Levo 400µg and Levo 200µg
Started | 11 | 12 | 12 | 12 | 13 | 12
Completed | 11 | 12 | 12 | 12 | 13 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (7 Days)
Arm/Group | Sequence 1: Levo 200 µg, Levo 400µg, Placebo | Sequence 2: Levo 400µg, Placebo and Levo 200µg | Sequence 3: Placebo, Levo 200µg and Levo 400µg | Sequence 4: Levo 200µg, Placebo, and Levo 400µg | Sequence 5: Levo 400µg, Levo 200µg and Placebo | Sequence 6: Placebo, Levo 400µg and Levo 200µg
Started | 11 | 12 | 12 | 12 | 13 | 12
Completed | 11 | 12 | 12 | 12 | 13 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Levocabastine: Participants received placebo/ Levo at a dose of 200 µg OD in the morning as 2 nasal sprays (50 µg per spray) into each nostril or 400 µg BID in the morning and evening as 2 nasal sprays (50 µg per spray) into each nostril for 7 days each, in a crossover design. Treatment was given in one of six sequences in Periods 1, 2, and 3, (14 to 20 day washout period between treatments): ABC, BCA, CAB, ACB, BAC, CBA (A, Levo 200µg; B, Levo 400µg: C, Placebo). On Day 8 of each treatment period (approximately 12 hours post dosing for treatment A and 24 hours post dosing for treatment B and C), participants entered the environmental exposure chamber (EEC) for a 4-hour period, and the assessments were conducted 12-24 hours post-dose. All participants attended a follow-up visit within 7 to 14 day after their final dose, and the overall duration for participation in the study (screening to follow-up) was 13 weeks.
Arm/Group | Placebo/Levocabastine
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 45
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 26
  Asian - Central/South Asian Heritage | 7
  Asian - East Asian Heritage | 3
  Asian - South East Asian Heritage | 3
  Asian - Mixed Race | 1
  White - Arabic/North African Heritage | 3
  White - White/Caucasian/European Heritage | 35

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean of the Total Nasal Symptom Score (TNSS) (0-4) Hours (h) Post Start of Allergen Chamber Challenge on Day 8
Description: The TNSS (score of 0-12) is defined as the sum of the symptom scores for the four individual components (nasal congestion, rhinorrhea, nasal itch, and sneezing, each scored on 0-3 scale [0=none, 1=mild, 2=moderate, 3=severe]). TNSS was measured at the pre-allergen chamber challenge, and then every 15 minutes from 0 to 4 hours post start of the allergen chamber challenge. In the Environmental Exposure Chamber (EEC), aerosolized allergen was administered in a sealed chamber to evaluate the efficacy of antihistamines/other treatments. Weighted mean TNSS was calculated by dividing the value of the area under the response time curve over the 0-4 hours (calculated by trapezoidal rule) by the time interval of available data.
Time Frame: Day 8 of each treatment period (up to 13 Weeks)
Population: Per Protocol Population: all participants in the Intent-to-Treat Population (defined as all participants who were randomized and received >= 1 dose of study medication) and not identified as full protocol deviators with respect to criteria that were considered to impact the primary efficacy analysis. Only those participants contributing data at the
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Placebo: Participants received placebo BID as 2 nasal sprays per nostril in the morning and evening for 7 days during one of three treatment periods. Each treatment period was followed by a washout period of 14 to 20 days.
- Levocabastine 200µg OD: Participants received levocabastine 200 µg once daily OD as two 50 µg nasal sprays into each nostril in the morning for 7 days during one of the three treatment periods. Each treatment period was followed by a washout period of 14 to 20 days.
- Levocabastine 400µg BID: Participants received levocabastine 400 µg BID as two 50 µg nasal sprays into each nostril in the morning and evening for 7 days during one of the three treatment periods. Each treatment period was followed by a washout period of 14 to 20 days.
Arm/Group | Placebo | Levocabastine 200µg OD | Levocabastine 400µg BID
Number analyzed (Participants) | 71 | 71 | 71
Scores on a scale | 5.190 [4.620 to 5.760] | 4.071 [3.502 to 4.641] | 3.840 [3.271 to 4.410]
Statistical Analysis 1: Comparison: Placebo vs Levocabastine 400µg BID; Test type: Superiority or Other; p < 0.0001, Mixed Model ANOVA; Mean Difference (Final Values) = -1.350, 95% CI 2-sided [-1.943 to -0.756]
Statistical Analysis 2: Comparison: Placebo vs Levocabastine 200µg OD; Test type: Superiority or Other; p = 0.0003, Mixed Model ANOVA; Mean Difference (Final Values) = -1.118, 95% CI 2-sided [-1.712 to -0.525]
Statistical Analysis 3: Comparison: Placebo vs Levocabastine 200µg OD vs Levocabastine 400µg BID; Test type: Non-Inferiority or Equivalence — Levocabastine OD would be declared as non-inferior to levocabastine BID if upper limit of 95% confidence interval of the treatment difference estimate (OD vs BD) was less than 1; Mean Difference (Final Values) = 0.231, 95% CI 2-sided [-0.361 to 0.823]

2. Secondary Outcome: Weighted Mean of the Symptom Scores for the Four Individual Components of the Total Nasal Symptom Score (TNSS) (Nasal Congestion, Rhinorrhea, Nasal Itching and Sneezing) (0-4) Hours Post Start of the Allergen Chamber Challenge on Day 8
Description: TNSS contains symtom scores for the four individual components (nasal congestion [NACG], rhinorrhea [RHSCR], nasal itching [NAITS] and sneezing [SNZS]), each scored on a 0 - 3 scale [0=none, 1=mild, 2=moderate, 3=severe]). TNSS was measured at the pre-allergen chamber challenge, and then every 15 minutes from 0 to 4 hours post start of the allergen chamber challenge. In the Environmental Exposure Chamber (EEC), aerosolized allergen is administered in a sealed chamber to evaluate the efficacy of antihistamines/other treatments. The participants recorded their symptom scores on an e-diary. The mean score for each participant was calculated using the available diary data from the assessment periods, taking the average of non-missing data during the period. Weighted mean of the individual symptoms of theTNSS were calculated by dividing the value of the area under the response time curve over the 0-4 hours (calculated by trapezoidal rule) by the time interval of available data.
Time Frame: Day 8 of each treatment period (up to 13 Weeks)
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Levocabastine 200µg OD | Levocabastine 400µg BID
Number analyzed (Participants) | 74 | 73 | 73
Scores on a scale
  NACG | 1.483 [1.322 to 1.643] | 1.217 [1.056 to 1.378] | 1.226 [1.065 to 1.387]
  RHSCR | 1.403 [1.232 to 1.574] | 1.035 [0.863 to 1.206] | 1.004 [0.833 to 1.176]
  NAITS | 1.257 [1.092 to 1.423] | 1.099 [0.932 to 1.265] | 1.040 [0.874 to 1.207]
  SNZS | 1.018 [0.857 to 1.178] | 0.647 [0.486 to 0.808] | 0.529 [0.368 to 0.690]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment until the follow-up contact (up to 13 weeks).
Description: SAEs and non-serious AEs were collected in members of the ITT Population, comprised of all randomized participants who received at least one dose of investigational product , according to the actual treatment received.
Arm/Group | Placebo | Levocabastine 200µg OD | Levocabastine 400µg BID
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/76 | 0/74
Other Adverse Events (participants affected / at risk) | 2/75 | 3/76 | 5/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | Levocabastine 200µg OD (N=76) | Levocabastine 400µg BID (N=74)
Headache (Nervous system disorders) | 1 | 0 | 3
Somnolence (Nervous system disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.